CLINICAL TRIAL: NCT06628687
Title: A Post-marketing, Observational, Descriptive Study to Assess the Risk Associated With Pregnancy, the Maternal Complications, and Adverse Effects on the Developing Fetus, Neonate, and Infant Among Individuals Exposed to Omaveloxolone During Pregnancy and/or Lactation
Brief Title: A Study to Learn How BIIB141 (Omaveloxolone) Affects the Health of Participants With Friedrich's Ataxia Who Took it During Pregnancy and/or During Breastfeeding and About the Health of Their Babies
Status: Recruiting | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 296FA402; EUPAS1000000327 (Other: EU PAS number)
Record Dates: First submitted 2024-09-30; First posted 2024-10-08 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — omaveloxolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Omaveloxolone: Participants with FA who were exposed to omaveloxolone at any time during pregnancy (from 12 days prior to conception through the end of pregnancy outcome), and/or at any time during lactation (up to 1 year of infant age or weaning, whichever comes first).
  Interventions: Drug: Omaveloxolone

INTERVENTIONS:
Drug: Omaveloxolone — Administered as specified in the treatment arm.
  Other Names: SKYCLARYS; BIIB141; RTA 408

SUMMARY:
In this study, researchers will learn more about the safety of BIIB141, also known as omaveloxolone or SKYCLARYS. This is a drug available for doctors to prescribe for people with Friedrich's Ataxia, also known as FA. This is known as an "observational" study, which collects health information about study participants without changing their medical care. Participants for this study will have taken BIIB141 at any time during pregnancy and/or while breastfeeding or pumping up through the first year after delivery. Participants can join this study on their own or they may be enrolled by their regular doctors. This study is also known as the "SKYCLARYS (Omaveloxolone) Pregnancy and Lactation Surveillance Program."

The main objective of this study is to learn more about how BIIB141 may affect pregnancy, as well as any effects on the health of the mother and of the baby during its first year of life.

The main question researchers want to answer in this study is:

· Does taking BIIB141 during pregnancy or breastfeeding lead to any major birth defects?

Researchers will also learn more about:

* Does taking BIIB141 during pregnancy or breastfeeding lead to any minor birth defects?
* Does taking BIIB141 during pregnancy or breastfeeding affect the following:
* Gestational diabetes, a disease that can happen during pregnancy that affects how your body uses sugar
* Pre-eclampsia, a pregnancy-related high blood pressure disease
* Unborn baby being small for its expected age (usually in weeks)
* Loss of an unborn baby
* Live birth
* Premature birth
* Loss of a newborn
* Growth or developmental delays in the baby
* Serious illness in the baby resulting in hospitalization
* Serious infections in the baby, or ones in babies with a weakened immune system

This study will be done as follows:

* Participants will join the study after signing an informed consent form, also known as an ICF.
* During the study, health information from the participants' regular visits to their doctor will be collected based on whether participant joined the study while pregnant or after the baby is born.
* Each participant will be in the study for up to 1 year after the birth of their child, unless they decide to leave early. Overall, this study is expected to last at least 10 years.

DETAILED DESCRIPTION:
The objective is to conduct a worldwide descriptive study to collect prospective and retrospective data in women exposed to omaveloxolone during pregnancy and/or lactation to assess risk associated with pregnancy, the maternal complications, and adverse effects on the developing fetus, neonate, and infant (through at least the first year of life) in the post-marketing setting.

ELIGIBILITY:
Key Inclusion Criteria:

- Exposure to omaveloxolone for FA at any time during pregnancy (from 12 days prior to conception to pregnancy outcome) and/or at any time during lactation (up to 1 year of infant age or weaning, whichever comes first).

Key Exclusion Criteria:

- Not having exposure to omaveloxolone for FA.

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The study population will include participants with FA who were exposed to omaveloxolone at any time during pregnancy and/or lactation.
  Participants will be enrolled prospectively and retrospectively. Women who enroll prior to pregnancy outcome, and/or prior to start of breastfeeding will be enrolled as prospective participants. Women who enroll after the pregnancy has occurred and/or following the start of breastfeeding will be enrolled as retrospective participants. Retrospective participants will not be included in the analysis population. For prospective and retrospective participants exposed during lactation only, data will be reported separately from pregnancy exposure cases.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-10-26 (Estimated); Primary Completion 2035-04-30 (Estimated); Study Completion 2035-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of Major Congenital Malformations (MCMs) | Up to 10 years
  A MCM is defined as an abnormality of body structure or function that is present at birth; is of prenatal origin (i.e., birth defect); has significant medical, social, or cosmetic consequences for the affected participant; and typically requires medical intervention.

SECONDARY OUTCOMES:
Number of Minor Congenital Malformations | Up to 10 years
  Minor congenital malformations include an anomaly or abnormality of body structure that is present at birth, is of prenatal origin (i.e., birth defect), poses no significant health problem in the neonatal period, and tends to have limited social or cosmetic consequences for the affected participant.
Number of Participants With Gestational Diabetes | Up to 9 months
Number of Participants With Pre-eclampsia | Up to 9 months
Number of Fetal Loss | Up to 9 months
  A fetal loss that occurs for any reason at any time during pregnancy will be reported.
Number of Spontaneous Abortions | Up to 9 months
  Spontaneous abortion refers to an involuntary fetal loss or the expulsion of the products of conception occurring prior to 20 gestational weeks.
Number of Stillbirths | Up to 9 months
  Still birth refers to an involuntary fetal loss occurring at or after 20 gestational weeks or, if gestational age is unknown, a fetus weighing ≥ 350 grams (g).
Number of Elective or Therapeutic Abortion | Up to 9 months
  Elective or therapeutic abortion refers to a voluntary fetal loss or interruption of pregnancy that occurs for any reason, including but not limited to for the preservation of maternal health or due to fetal abnormalities.
Number of Live Births | Up to 9 months
  Live birth refers to the birth of a living fetus after 20 weeks of gestation or, if gestational age is unknown, weighing ≥ 350 g.
Number of Preterm Births | Up to 9 months
  Preterm birth refers to a live birth at or before 37 weeks of gestation.
Number of Small for Gestational Age (SGA) | Up to 9 months
  SGA is defined as birth weight less than 10th percentile for sex and gestational age using standard growth charts for full and preterm live-born infants.
Number of Neonatal Deaths | Within 28 days postdelivery
  Neonatal death refers to the death of a live-born infant within the first 28 days of life.
Number of Infant Deaths | Up to approximately 1 year
  Infant death refers to the death of a live-born infant within the first year of life.
Number of Infants with Abnormal Postnatal Growth and Development | Up to approximately 1 year
  Infant growth measurements will be used to estimate gender-specific weight-for-length, head circumference-for-age, length-for-age, and weight-for-age percentiles. Developmental milestones (i.e., social/emotional, language/communication, neurocognitive, movement/physical development) will be evaluated to determine results of infant status (i.e., infants who are failing to achieve at least one milestone in any category will be considered developmentally delayed in that category).
Number of Infant Hospitalization due to Serious Illness | Up to 1 year
  Infant hospital visit due to a serious (that is, results in significant disability, incapacity, or death; is life-threatening; requires inpatient or prolonged hospitalization; or is considered medically important) illness will be reported.
Number of Infant Serious or Opportunistic Infections | Up to 1 year
  Infections that occur within an infant's first year of life and is either opportunistic (i.e., occurs more often or is more severe in people with weakened immune systems than in people with healthy immune systems) or serious (that is, results in significant disability, incapacity, or death; is life-threatening; requires inpatient or prolonged hospitalization; or is considered medically important) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Evidera, Morrisville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/